CLINICAL TRIAL: NCT07342738
Title: A Cliniacl Study of T Cell Receptor-engineered T-Cell (TCR-T) Injection in Patients With Advanced Solid Tumors Induced by Kirsten Rat Sarcoma Viral Oncogene Homolog (KRAS) Mutations.
Brief Title: TCR-T Cell Therapy for KRAS Mutation in Advanced Solid Tumors
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: Shanghai Bintie Biotechnology Co., Ltd (Unknown)
Responsible Party: Principal Investigator, Yuhong Li, MD, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BT004 TCR-T
Record Dates: First submitted 2026-01-05; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: KRAS G12V; KRAS G12D; Solid Tumor
MeSH Terms: interventions — fludarabine; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TCR-T cells (Experimental): TCR-T cells targeted for KRAS mutation
  Interventions: Biological: TCR-T cells; Drug: Fludarabine; Drug: Cyclophosphamide

INTERVENTIONS:
Biological: TCR-T cells — TCR-T cell injection will be administered intravenously after lymphodepletion.
Drug: Fludarabine — Fludarabine is used for lymphodepletion.
Drug: Cyclophosphamide — Cyclophosphamide is used for lymphodepletion.

SUMMARY:
This is a single-arm, Multicenter, open-label clinical study aimed at evaluating the safety and efficacy of TCR-T injection in patients with advanced solid tumors induced by KRAS mutations.

DETAILED DESCRIPTION:
This study is planned to enroll patients with advanced solid tumors who have KRAS G12V or G12D mutations and matching Human Leukocyte Antigen(HLA)-A*11:01 or HLA-C*01:02 subtypes. The study consists of screening period, leukapheresis period, lymphodepletion period, treatment period, observation period and follow-up period. The patients were treated lymphodepletion treatment with cyclophosphamide and fludarabine and than infused TCR-T. All subjects who have received TCR-T injection will be followed for safety and efficacy up to 1 years.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary signing of an informed consent form (ICF)；
2. Males or females, aged 18-70 years (inclusive);
3. Subjects with advanced solid tumors confirmed by histology/cytology, have failed with standard treatment, or intolerant to standard treatment, or no standard treatment exists：1）Colorectal cancer：failed or intolerant to at least two lines of standard treatment.2）Non-small cell lung cancer：Absence of the following gene mutations (Epidermal Growth Factor Receptor[EGFR]、Anaplastic Lymphoma Kinase[ALK] 、 Proto-oncogene tyrosine-protein kinase 1[ROS1]) and having failed or intolerant to platinum-based chemotherapy and/or immunotherapy and/or anti-angiogenic therapy.3）Other advanced solid tumors：failed with standard treatment, or intolerant to standard treatment, or no standard treatment exist.
4. At least one measurable lesion (according to Response Evaluation Criteria in Solid Tumors[RECIST], version 1.1);
5. Patients with tumor tissue or peripheral blood testing positive for KRAS-G12V or G12D mutations and expression of matching HLA-A*11:01 or HLA-C*01:02 subtypes;
6. ECOG (Eastern Cooperative Oncology Group)≤2;
7. Life expectancy ≥3 months;
8. Adequate functional reserve of organs：1）Hematology (no intensive blood transfusion, platelet transfusion or cell growth factor performed within 14 days before the test)：·Absolute neutrophil count ≥1×10E9/L;·Platelet count ≥50×10E9/L, hemoglobin>90g/L;·Absolute lymphocyte count ≥0.5×10E9/L;2）Blood chemistry：·Alanine aminotransferase (ALT) ≤3×Upper Limit of Normal (ULN);·Aspartate aminotransferase (AST) ≤3×ULN（patients with hepatic metastasis, ALT and AST ≤5×ULN）;·Serum creatinine ≤1.5×ULN or Creatinine clearance ≥50 mL/min;·Total bilirubin (TB) ≤1.5×ULN；3）Blood chemistry：·APTT≤1.5×ULN，INR≤1.5×ULN4）The subject has left ventricular ejection fraction (LVEF) ≥ 50% and no clinically significant pericardial effusion diagnosed by echocardiography;5）No clinically significant electrocardiographic abnormality;6）Basic oxygen saturation is >92% under the indoor natural air environment.
9. Women of childbearing age must be negative for blood HCG (Human Chorionic Gonadotropin) pregnancy test (by immunofluorescence method) at screening and baseline periods, and agree to use effective contraception for at least 1 year after infusion; and male subjects whose partners are women of childbearing age must agree to use effective barrier contraception methods and avoid sperm donation for at least 1 year after infusion.

Exclusion Criteria:

1. Other malignancies (except non-melanoma skin cancer with the disease-free survival of more than 5 years and cervical carcinoma in situ, bladder cancer, or breast cancer);
2. History of organ transplantation；
3. A history of mental disorders, which may affect compliance with this protocol or lead to failure in signing the ICF;
4. A history of autoimmune diseases (e.g., Crohn's disease, rheumatoid arthritis and systemic lupus erythematosus) requiring systemic immunosuppressive/systemic disease-modulating drugs；
5. Poorly controlled hypertension with drug (systolic blood pressure >160 mmHg and/or diastolic blood pressure >100 mmHg) or occurrence of grade III-IV heart failure or myocardial infarction, cardiac angioplasty or stent placement, unstable angina pectoris, or other clinically significant heart diseases within one year prior to signing the ICF; Corrected QT Interval (QTc) interval >450 ms for males or QTc interval >470 ms for females during screening (QTc interval calculated using the Fridericia formula)；
6. Patients with intestinal obstruction or obstructive jaundice and are deemed ineligible for enrollment by the investigator；
7. Symptomatic intracranial metastases, or moderate to severe ascites or pleural effusion requiring drainage to relieve symptoms；
8. A history of or any central nervous system disorders, such as epileptic seizure, cerebrovascular ischemia/hemorrhage, dementia, cerebellar disease, or any autoimmune disease involving the central nervous system within the past 6 months；
9. A positive result obtained in any of the following virological tests:1）Antibody to human immunodeficiency virus (HIV antibody); 2）Hepatitis C virus antibody (HCV antibody), with a positive result for hepatitis C virus ribonucleic acid (HCV RNA); 3）Positive for hepatitis B surface antigen (HBsAg); or positive for hepatitis B core antibody (HBcAb) and positive for hepatitis B virus deoxyribonucleic acid (HBV DNA) copies ≥2000 IU/mL; 4）Treponema pallidum antibody (TP antibody) and positive for unheated serum reagin test;
10. Fungal, bacterial, viral or other infections or suspected fungal, bacterial, viral or other infections that cannot be controlled or require intravenous administration；
11. Significant tendency for bleeding, such as active gastrointestinal bleeding, coagulation disorders；
12. Deep vein thrombosis requiring treatment within the past 6 months, unless the risk of thrombosis is acceptable after treatment, as assessed by the investigator；
13. Interstitial lung disease (such as interstitial pneumonia, pulmonary fibrosis), or a history of clinically significant respiratory system diseases at screening；
14. Use of granulocyte colony-stimulating factor (G-CSF) or granulocyte-macrophage colony-stimulating factor (GM-CSF) within 2 weeks prior to leukapheresis；
15. Participation in any other clinical studies within 1 month prior to signing the master informed consent form；
16. Patients with poor compliance due to physiological, family, social, geographic and other factors, and failure to follow the study protocol and the follow-up plan；
17. Patients with contraindications to drugs used in the study；
18. Comorbidities requiring treatment with systemic corticosteroids (dexamethasone at a dose of ≥ 5 mg/day or other corticosteroids at the equivalent dose) or other immunosuppressive drugs after initiation of the study treatment, as judged by the investigator；
19. Women who are breastfeeding and are unwilling to stop breastfeeding；
20. Any other conditions that are, in the opinion of the investigator, not suitable for enrollment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2028-02-01 (Estimated); Study Completion 2029-02-01 (Estimated)

PRIMARY OUTCOMES:
Adverse Events (AEs) | 1 year
  Incidence and severity of adverse events
Serious Adverse Events (SAEs) | 1 year
  Incidence and severity of serious adverse events

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | 1 year
  The percentage of participants who achieved Complete Response (CR) or Partial Response (PR) based on RECIST version 1.1
Disease Control Rate (DCR) | 1 year
  The percentage of participants who achieved Complete Response (CR) or Partial Response (PR) or Stable disease (SD) based on RECIST version 1.1
Duration of response (DOR) | 1 year
  DOR is defined as the time from the first evaluation of a tumor as CR or PR to the first evaluation as progressive disease (PD) or death from any cause
Time to response (TTR) | 1 year
  TTR is defined as the time between cell infusion and initial disease assessment as CR or PR
Progression-free survival (PFS) | 1 year
  PFS is defined as the time from the date of cell infusion until the date of tumor progression or death from any cause
Overall survival (OS) | 1 year
  OS is defined as the time between the date of cell infusion and the death of the patient for any reason
Cmax of TCR-T cells after infusion | 1 year
  Peak peripheral blood concentration of TCR-T cells following infusion, measured by flow cytometry.
Tmax of TCR-T cells after infusion | 1 year
  Time to reach maximum observed concentration (Tmax) of TCR-T cells
Peak level of cytokines in serum after infusion | 1 year
  The cytokines mainly include interleukin-2 (IL-2 ), IL-6, IL-8, IL-10, tumor necrosis factor-α (TNF-α), C reactive protein (CRP),Interferon gamma (IFN-γ) .Peak was defined as the maximum post-baseline level of the cytokine.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No